CLINICAL TRIAL: NCT06429020
Title: Sonography for COVID-19 Vaccines Related Reactive Lymphadenopathy: A Retrospective Study
Brief Title: Sonography for COVID-19 Vaccines Related Reactive Lymphadenopathy
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMMC11201-010
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Reactive Axillary Lymphadenopathy for SARS-CoV-2 Vaccines in the Asian Taiwanese Population
Keywords: Breast Neoplasms; covid-19 vaccine; lymphadenopathy
MeSH Terms: conditions — Breast Neoplasms; Lymphadenopathy | interventions — Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: non SARS-COV-2 vaccinated group
- vaccinated group: SARS-COV-2 vaccinated group
  Interventions: Biological: the AstraZeneca ChAdOx1 (AZ) vaccine, Moderna mRNA-1273 (Moderna) vaccine, and Pfizer-BioNTech BNT162b2 (BNT) vaccine.

INTERVENTIONS:
Biological: the AstraZeneca ChAdOx1 (AZ) vaccine, Moderna mRNA-1273 (Moderna) vaccine, and Pfizer-BioNTech BNT162b2 (BNT) vaccine. — record the condition of vaccination
  Groups: vaccinated group

SUMMARY:
This study aimed to provide vast clinical information to facilitate breast sonographic examination for participants who underwent recent SARS-CoV-2 vaccination.

Among different SARS-CoV-2 vaccines in the Asian Taiwanese population, reactive axillary lymphadenopathy was investigated through breast sonographic findings and clinical data analysis. The sample included participants with recent vaccinations by different brands approved in Taiwan.

DETAILED DESCRIPTION:
Study Design and Sample The retrospective study included female patients who underwent breast sonography in the radiology department of Chi Mei Medical Center between July 2021 and March 2022. The patients' breast cancer history and COVID-19 vaccination history were collected and analyzed.

Analysis of Breast Sonography Lymphadenopathy is defined as an enlarged lymph node with cortical thickening >3 mm, either concentric or eccentric, with or without effacement of fatty hilum, or in-creased non-hilar vascularity on color or power Doppler. The positive axillary lymph node findings were correlated by confirming a link to SARS-CoV-2 vaccination history within 90 days in the ipsilateral arm.

Statistical Analysis All statistical analyses were performed using the R Stats package. Descriptive summaries were reported as mean ± standard deviation for continuous variables and percentages for categorical variables. For non-parametric variables, median with interquartile range and Mann-Whitney U test were used. Statistical significance was set at a p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* female patients receiving breast sonography

Exclusion Criteria:

* receive Covid 19 vaccine other than AZ, BNT, Moderna
* Ongoing primary breast malignancy
* History of malignancy other than primary breast malignancy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent breast sonography in the radiology department of Chi Mei Medical Center between July 2021 and March 2022.
Sampling Method: Probability Sample
Enrollment: 1089 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Presentation of axillary lymphadenopathy in sonographic examination | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pin Chi Huang, Study Chair — ChiMei Medical Center, Taiwan, R.O.C.
Locations (1):
- ChiMei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No